CLINICAL TRIAL: NCT01611402
Title: Transcriptional Signature of HIV And TB Co-Infection
Brief Title: Gene Expression in HIV and Tuberculosis Co-infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120142; 12-I-0142
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-04-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; HIV Infection; Transcriptional Signature; IRIS
MeSH Terms: conditions — Tuberculosis; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Tuberculosis (TB) infection is particularly deadly when it happens in people who are also infected with the human immunodeficiency virus (HIV). However, not much is known about how these two infections affect each other. Some people who have HIV or TB infections develop health problems after they start taking either HIV or TB medications or both. These drugs can improve the body s ability to fight infections, but sometimes this sudden improvement can make the infected person initially become sicker. Researchers want to study how these infections affect the immune system and the gene expression of people who have TB and may or may not have HIV, to see if there is a pattern of gene expression that may predict whether people starting treatment may get sicker initially.

Objectives:

- To study the gene expression and immune systems of people with TB who may or may not also have HIV.

Eligibility:

* Adults at least 18 years of age who have tuberculosis.
* Participants will be drawn from study sites in the United States and China.

Design:

* Participants will be divided into three study groups. The first group will have TB but not HIV. The second group will have both TB and HIV that have not been treated. The third group will have both TB and HIV that are currently being treated.
* All participants will have a single study visit. Blood samples will be collected at this visit. A medical history will also be collected.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains one of the deadliest infections throughout the world, particularly in the setting of HIV infection. In China, TB is a frequently diagnosed complication of HIV infection. The immunopathogenesis of TB remains unclear, and although it is known that HIV infection increases the risk of developing active TB, either through infection or reactivation of latent disease, how it does so has yet to be determined. It is also known that patients co-infected with HIV and TB and na(SqrRoot) ve to antiretroviral therapy (ART) have a particularly high risk of developing Immune Reconstitution Inflammatory Syndrome (IRIS) after ART therapy is initiated, but the immunopathogenesis of this reaction is also unclear.

The use of genomics has significantly improved the understanding of disease pathogenesis and is increasingly being used to predict responses to therapy as well. Recently, blood transcriptional signatures capable of distinguishing active and latent TB infection have been identified using highly parallelized analytical platforms capable of simultaneous survey of transcription of known genes. These signatures have hinted at a complex role for type I interferons in the development of active TB infection, but this has not yet been studied in people with HIV and TB co-infection. Further in depth studies are needed to characterize the spectrum of responses to TB/HIV co-infection, and how these responses correlate with clinical data.

We propose a cross-sectional cohort study, to be conducted in both the US and in China, to identify blood mRNA expression profiles distinguishing TB mono-infected and TB/HIV co-infected ART-na(SqrRoot) ve patients from treated patients with and without TB-IRIS. Secondary objectives will include correlating gene expression levels with clinical outcomes and soluble biomarkers. The study will comprise a test set (in China) of up to 140 patients divided among the different cohorts and a validation set (in the US) of up to 125 patients divided among the three groups Participation will involve a single study visit to consist of small volume phlebotomy (approximately 25 mL for safety labs, transcriptome analysis, lymphocyte counts, and serum and plasma storage) a urine sample and information gleaned from the clinical record entered into a coded Case Report Form (CRF). The U.S. cohort will have an additional 40 mLs of blood collected for mononuclear cells (total of approximately 65mLs).The study will exclude women who are pregnant or breast-feeding (which can be associated with immune compromise and changes in markers associated with inflammation), and persons with anemia (who may be unable to tolerate phlebotomy solely for research purposes).

ELIGIBILITY:
* INCLUSION CRITERIA:

For all patients:

* Adults, age 18 or older
* TB diagnosis, ascertained as follows:

  1. specimen or biopsy smear, culture, or PCR positivity or
  2. compatible clinical presentation and imaging with strong suspicion for TB that necessitates initiation of empiric TB therapy (in which case the confirmation by culture or other laboratory means may follow enrollment, or alternatively clinical improvement in response to TB therapy may confirm the diagnosis).

If the TB diagnosis cannot be confirmed as above (i.e. culture positive for NTM), the patient will be excluded from final analysis.

* Ability and willingness of subject or legal guardian/representative to understand study requirements and give informed consent. In the event an adult subject is unable, due to illness or mental incapacity, to give informed consent, a person authorized with durable power of attorney (DPA) or legal guardian may give consent for the subject s blood to be obtained, shipped, and tested under this protocol.
* Agree to storage of study data and biologic specimens for use in future studies of immune function, tuberculosis, genetics, and/or HIV pathogenesis.

Patients in TB mono-infected arm (Group A) would additionally be eligible if:

* HIV negative (documented seronegative within 1 month of study visit)
* Not receiving TB therapy for more than 7 days prior to study visit (Group A1) or
* Currently on TB therapy for >7 days and < 5 months (Group A2)

Patients in TB/HIV co-infected arm (Group B) would additionally be eligible if:

* HIV positive (outside HIV testing will be accepted)
* Not receiving TB therapy for more than 7 days prior to study visit
* Untreated or ART na(SqrRoot) ve (will be accepted if they had been on ART in the past but none within the last 6 months).

Patients in TB/HIV co-infected, treated arm (Group C) would additionally be eligible if:

* HIV positive
* Currently receiving TB therapy
* Currently receiving ART (The subset of patients without TB-IRIS will have been on antiretroviral therapy for at least 8 and not more than 12 weeks. The subset of patients with TB-IRIS will be enrolled at the time of their TB-IRIS event) with some evidence of adherence (often measured by clinical improvement, medication refills or laboratory values)
* The TB-IRIS subset of patients (15 patients at NIAID and 20 patients at SHAPHC) would also need to meet criteria for paradoxical TB-IRIS

EXCLUSION CRITERIA:

Pregnancy or post-partum period (6 months post-partum or while breast-feeding, whichever is longer).

Documented history of hemoglobin from most recent blood draw less than 7g/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-05-29; Study Completion 2016-04-06

PRIMARY OUTCOMES:
Identify blood mRNA expression profiles distinguishing TB onoinfectedfrom TB/HIV co-infected patients (ART-naive and ART-treated with and without TB-IRIS). | During data analysis phase

SECONDARY OUTCOMES:
Correlate gene expression levels with clinical and laboratory variablesincluding flow cytometry and soluble biomarkers. | During data analysis phase
Quantify the tuberculosis antigen load at the beginning of anti-TB therapy by lateral flow lipo-arabinomannan assay (TB-LAM LFA) and study how the antigen burden affects the disease presentation (including radiographic findings), or transcriptio... | During data analysis phase.
Study separated cell populations (monocytes, dendritic cells, NK, T cell subsets or neurtrophils) to validate any identified transcriptional signature or to further investigate pathogen-specific responses. | During data analysis phase

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Meintjes G, Rabie H, Wilkinson RJ, Cotton MF. Tuberculosis-associated immune reconstitution inflammatory syndrome and unmasking of tuberculosis by antiretroviral therapy. Clin Chest Med. 2009 Dec;30(4):797-810, x. doi: 10.1016/j.ccm.2009.08.013. PMID 19925968
- [Background] Harries AD, Zachariah R, Corbett EL, Lawn SD, Santos-Filho ET, Chimzizi R, Harrington M, Maher D, Williams BG, De Cock KM. The HIV-associated tuberculosis epidemic--when will we act? Lancet. 2010 May 29;375(9729):1906-19. doi: 10.1016/S0140-6736(10)60409-6. Epub 2010 May 18. PMID 20488516
- [Background] Houben RM, Crampin AC, Ndhlovu R, Sonnenberg P, Godfrey-Faussett P, Haas WH, Engelmann G, Lombard CJ, Wilkinson D, Bruchfeld J, Lockman S, Tappero J, Glynn JR. Human immunodeficiency virus associated tuberculosis more often due to recent infection than reactivation of latent infection. Int J Tuberc Lung Dis. 2011 Jan;15(1):24-31. PMID 21276292